CLINICAL TRIAL: NCT03548363
Title: A Double-blind, Randomized, Placebo-controlled Clinical Study to Evaluate the Efficacy of Gingest on Symptoms of Dyspepsia
Brief Title: Effect of Gingest on Symptoms of Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantia Food Clinical Trials (Industry)
Collaborators: Givaudan France Naturals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFCRO 085
Record Dates: First submitted 2018-04-11; First posted 2018-06-07 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Dyspepsia; Epigastric Fullness; Bloating; Epigastric Pain
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, 4-week parallel intervention in subjects with mild to moderate Dyspepsia (as defined by the Leeds Dyspepsia Questionnaire) in 3-treatment arms: 1.) 100 mg/d Gingest; 2.) 200 mg/d Gingest; 3.) Placebo (maltodextrin)
Who Masked: Participant, Investigator
Masking Description: Both the investigators with any involvement in the study or data analysis prior to database locking and subjects are blinded to what treatment they receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gingest High (Active Comparator): 200 mg/d Gingest (powdered extract obtained from Ginger rhizomes) for 4-weeks
  Interventions: Dietary Supplement: Gingest powdered extract obtained from Ginger rhizomes
- Gingest low (Active Comparator): 100 mg/d Gingest (powdered extract obtained from Ginger rhizomes) + 100 mg maltodextrin for 4-weeks
  Interventions: Dietary Supplement: Gingest powdered extract obtained from Ginger rhizomes
- Placebo (Placebo Comparator): 200 mg/d maltodextrin for 4-weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Gingest powdered extract obtained from Ginger rhizomes — Description: Powdered extract obtained from Ginger rhizomes. Botanical name: Zingiber officinale Roscoe Plant part used: Dried rhyzome Extraction solvent: CO2 Extract Ratio 45-60 / 1 100mg of extract are equivalent to an average of 4400 mg of dry ginger rhizomes
  Composition: Natural extract, Calcium Hydroxide, Polysorbate 80, De-oiled soya lecithin, Calcium silicate
  Arms: Gingest High; Gingest low
Dietary Supplement: Placebo — 200 mg/d maltodextrin
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, placebo controlled study on the effect of Gingest (ginger root extract) on symptoms of dyspepsia in 150 participants with mild to moderate dyspepsia.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is a chronic disorder of sensation and movement (peristalsis) in the upper digestive tract. A diagnosis of functional dyspepsia is determined when there is no evidence of structural disease and there have been at least three months of one or more of the following (with onset at least six months earlier). Ginger (Zingiber officinale) is traditionally used to treat a number of medical conditions, including those affecting the digestive tract, such as dyspepsia, flatulence, nausea and abdominal pain. Recent human clinical studies have found beneficial effects of ginger extract in patients with dyspepsia and gastric emptying in healthy populations.

The aim of the present study is therefore to investigate if two different doses of Gingest (100mg and 200 mg) reduces intensity of functional dyspepsia (based on a symptom severity questionnaire) compared to placebo (maltodextrin) in 150 subjects with mild to moderate dyspepsia (as determined through the Leeds Dyspepsia Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy free-living men and women,
2. Be aged 30 to 55 years (inclusive),
3. Be willing to provide informed consent,
4. Subject has upper abdominal pain or discomfort that is an unpleasant sensation, characterized by one or more of the following symptoms: early satiety, postprandial fullness, bloating, and nausea for at least 3 months during last year, without an identifiable underlying structural or biochemical motivation.
5. Leeds Dyspepsia Questionnaire score 8 to 24 (mild-moderate)
6. Beck's Depression Inventory score between 4 and 15

Exclusion Criteria:

1. Pregnancy/lactation
2. Subjects with relevant gastroesophageal reflux symptoms (retrosternal pain, burning, or regurgitation.
3. Subjects with clear evidence of irritable bowel syndrome.
4. Subjects under treatment with pharmacological substances that could influence the gastrointestinal system, such as prokinetics, ursodeoxycholic acid (UDCA), nonsteroidal anti-inflammatory drugs (NSAIDs), cholagogues, protonpump inhibitors, and H2 blockers, were asked to interrupt this treatment for one month before starting the study treatment.
5. Subjects with previous diagnosis of cancer or with previous surgery of the upper gastro gastrointestinal endoscopy were performed in order to exclude the presence of structural or biochemical causes of dyspepsia.
6. Participants are asked to avoid all foods containing ginger within the 14 days prior to study product administration and throughout the study. A list of foods high in ginger will be provided to subjects as a guide and this list will be reviewed at each visit.
7. Subject with known allergy to components of the test product
8. Any medical condition deemed exclusionary by the Principal Investigator
9. Subject has a history of drug and / or alcohol abuse at the time of enrolment
10. Change of dietary habit within the preceding month
11. Subject with known organic disease, including an inflammatory bowel disease, a benign or malign tumour of intestine or colon and significant systemic disease
12. Subject currently involved in any other clinical trial or having participated in a trial within the preceding 60 days,
13. Subject has any concurrent medical or psychiatric condition that, in the opinion of the Investigator, would compromise his/her ability to comply with the study requirements,
14. Current illnesses which could interfere with the study (e.g. prolonged severe diarrhea, regurgitation/severe, difficulty swallowing)
15. Subject has a history of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years,
16. Subject has a significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would preclude supplement ingestion and/or assessment of safety and the study objectives,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Intensity of functional dyspepsia symptom score over 4-weeks as measured by subject rating score at week-4 | 4-weeks
  Overall score indicates the intensity of functional dyspepsia as defined by Subject's rating after four weeks of intervention with Gingest (100mg and 200mgs) versus placebo. The lower the score, the higher the intensity of the dyspeptic symptoms.
  0: Not improved or worsened
  1. Slightly improved
  2. Markedly improved
  3. Completely improved

SECONDARY OUTCOMES:
Intensity of functional dyspepsia symptoms over 2-weeks as measured by subject rating score | 2-weeks
  Overall score indicates the intensity of functional dyspepsia as defined by Subject's rating after two weeks of intervention with Gingest (100mg and 200mgs) versus placebo.
  0: Not improved or worsened
  1. Slightly improved
  2. Markedly improved
  3. Completely improved
Severity of dyspeptic symptoms as measured by subject severity score measured at week-4. | 4-weeks
  Overall severity of specific suite of dyspeptic symptoms (including epigastric fullness, bloating, early satiety, nausea, vomiting epigastric pain) Absence of symptoms =0 Mild Symptoms = 1 Moderate Symptoms = 2 Severe symptoms = 3
Participant Global Assessment as measured by Participant Global Assessment Score at week-4 | 4 weeks
  Participant Global Assessment Short Form 36 assesses the overall general mental and physical health. Answers are combined to produce the following.
  Physical function score= a higher score means better health Role limitation due to physical health Score: a lower score means better health Role limitations due to emotional problems Score: a lower score means better health Energy/ fatigue Score: a lower score means better health Emotional well-being Score: a higher score means better health Social Functioning Score: a higher score means better health Pain Score: a lower score means better health General health Score: a higher score means better health
Leeds Dyspepsia Questionnaire as measured by total score at week-4 | 4 weeks
  Overall score is calculated from subject rating for frequency and severity responses for each symptom of dyspepsia.
  a summed total score of the frequency and severity responses for each symptom( Indigestion, heartburn, regurgitation, nausea combined) range: 0-32). 0= least severe.32= most severe each symptom = indigestion, regurgitation, heartburn and nausea a summed score of the frequency responses for each symptom (range: 0-16); a summed score of the severity responses for each symptom (range: 0-16); a categorized score of the single most frequent symptom (range: 0-4) and a categorized score of the single most severe symptom (range: 0-4).
Profile of Mood States Questionnaire (POMS) as measured by score at week-4. | 4 weeks
  Overall score assess changes in mood Not at all= 0 little = 1 Moderately = 2 Quite a lot = 3 Extremely = 4 Answers are combined. Higher the score for negative feelings i.e. tense the worse the mood. Higher the score for positive feelings i.e. Energetic the better the mood.
Beck's Depression Inventory as measured by score at week-4. | 4 weeks
  Overall score indicates severity of depressive symptoms
  1-10 = These ups and downs are considered normal 11-16__ Mild mood disturbance 17-20__Borderline clinical depression 21-30_Moderate depression 31-40_Severe depression over 40__________________Extreme depression
Cortisol awakening response (nmol/L) at week-4. | 4 weeks
  Measures salivary cortisol (nmol/L)
Reduction in medication to manage number of episodes requiring medication for dyspeptic symptoms as measured at week-4 | 4 weeks
  Number of times medication is taken to manage dyspeptic symptoms
Safety as assessed by adverse events and serious adverse events ongoing throughout the trial | 4 weeks
  Number of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia CRO, Heron House, Blackpool, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No
All data will remain proprietary and will only be shared with Naturex (commercial partner) and contract statisticians.